CLINICAL TRIAL: NCT05424328
Title: Virtual Planning Of Anterolateral Thigh Free Flap for Reconstruction Of Hemiglossectomy
Brief Title: Virtual Planning of ALT Flap
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Fellow left UF study never started
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202201118
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Tongue SCC
Keywords: SCC, Hemi glossectomy, ALT Flap. virtual planning

STUDY DESIGN:
Intervention Model Description: This study consists of 2 groups A and B each contains 10 patients of total 20 patients. Where group A (control group) where Alt flap harvest for tongue reconstruction after hemi glossectomy is done with the conventional method where flap design and volume depends on surgeon's own experience while group B (study group) the Alt flap design and volume will be harvested by the aid of a guide that is virtually planned before the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group: ALTF with preoperative virtual planning (Experimental): Subjects will receive ALTF( Anterolateral thigh flap) with preoperative virtual planning
  Interventions: Procedure: ALTF (Anterolateral thigh flap) with preoperative virtual planning
- Control Group: ALTF with conventional method (Active Comparator): Subjects will receive ALTF (Anterolateral thigh flap) with conventional method
  Interventions: Procedure: ALTF (Anterolateral thigh flap) with conventional method

INTERVENTIONS:
Procedure: ALTF (Anterolateral thigh flap) with preoperative virtual planning — In this study group, using preoperative CTs (head & neck and thigh ) to virtually plan a guide that can be used during the surgery, this guide will determine the design and dimensions of the Alt flap to be harvested and restore the defect left on the tongue due SCC resection and hemi glossectomy.
  Arms: Study Group: ALTF with preoperative virtual planning
Procedure: ALTF (Anterolateral thigh flap) with conventional method — ALTF (Anterolateral thigh flap) will be harvested with conventional method which depends on surgeon's own experience in determining the flap design and dimensions needed to reconstruct and restore the defect left on the tongue due SCC resection and hemi glossectomy.
  Arms: Control Group: ALTF with conventional method

SUMMARY:
This study evaluates the advantage of using preoperative virtual planning to design the volume and shape of antero-lateral thigh free flap tissue transfer to reconstruct tongue defects resulted from carcinoma resection and see how this would affect tongue form and speech function.

DETAILED DESCRIPTION:
This is a prospective randomized clinical study consisting of 2 groups A and B each contains 10 patients of total 20 patients. Where group A (control group) where Alt flap harvest for tongue reconstruction after hemi glossectomy is done with the conventional method while group B (study group) the Alt flap design and harvest is virtually planned before the operation.

The main issue regarding tongue reconstruction with ALTF is the matching of the size and shape between the harvested flap and the tongue defect assuming the hypothesis that an adequate flap volume is crucial for maintaining tongue function. Meanwhile, the preoperative planning of soft tissues is relatively difficult due to an undefined standardization and reference points. In this study, investigators will evaluate the use of preoperative virtual planning and 3D reconstructions for the restoration of tongue defects with ALTF. In this study, virtual surgical planning for the resection of the tongue cancer (hemi-glossectomy) will be used and will address flap design, which the investigators will base on anatomical landmarks using the preoperative virtual planning technology. The research team will compare the functional ( speech) and cosmetic outcomes of the virtually planned ALTF technique with the conventional method for hemi-glossectomy and reconstruction. The null hypothesis of this study is that there is no significant difference in functional & cosmetic outcome between the virtually planned ALTF technique with the conventional method for hemi-glossectomy and reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary tongue squamous cell carcinoma (SCC) requiring hemi-glossectomy.
2. No alveolar ridge involvement by the tumor process.
3. Planned to undergo tongue reconstruction using ALTF.
4. Patients with a depth of invasion more than 10mm but not crossing midline according to the classification of Ansarin et. al., we perform type IIIA glossectomy.

Exclusion Criteria:

1. Medically unfit patients; those who are not good candidates for long microvascular surgical reconstructive procedures e.g.: advanced Cardiopulmonary diseases.
2. Recurrent tongue carcinoma.
3. Patients with lesions invading the alveolar ridge.
4. Missing or non-compliance for imaging investigations.
5. Patients underwent preoperative adjuvant therapies.
6. No children will be involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Prospectively evaluate a new method of virtually planned ALTF and changes in flap volume for the reconstruction of tongue defects following hemi-glossectomy | Changes in flap volume/cm3 will be measured after one and six months after surgery where the preoperative virtually planned volume/cm3 is being the base line.
  Investigators will preoperatively use CT measurements and virtual planning 3D software to calculate the required ALT flap volume /cm3 by measuring flap dimensions (height, width and length) /cm3 and compare it with the postoperative real outcomes by re-measuring the real flap dimensions ( height, width and length) /cm3 .

SECONDARY OUTCOMES:
Assessment of Intelligibility of Dysarthric Speech (AIDS) test will be used to assess tongue speech functions following tongue reconstruction and compare speech changes. | Changes of speech will be compared After one and six months after surgery where the preoperative speech will be the base line.
  - In the AIDS test the speech analysist examiner will randomly select two sentences (5-15 words) for a total of 22 sentences utilizing table in manual, and reads them aloud once and then allow patients to say them while audio records each session via voice app on phone.
  Judge from the investigators will listen and transcribe. Making a report and develop outcomes.
  * Scoring will be according the standard scores of the AIDS test analysis where:
  * Intelligibility: Corresponds to number of correct words.
  * Speaking rate: Corresponds to words per minute (WPM) / duration of sentence samples in minutes
  * Rate of intelligible speech (intelligible words per minute (IWPM)): number of words identified correctly /total duration
  * Rate of unintelligible (unintelligible words per minute (UWPM)): number of unintelligible/total duration
  * Communication efficiency ratio: IWPM/190 IWPM.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Fernandes, MD, DMD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No